CLINICAL TRIAL: NCT06877702
Title: A Phase 1, 2-Part, Open-label Study to Evaluate Relative Bioavailability of Alternate Formulations of BMS-986460 in Healthy Adult Male Participants (Part 1), and a Single Ascending Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of BMS-986460 in Healthy Adult Male Participants (Part 2)
Brief Title: A Single-dose Study to Evaluate the Safety, Tolerability, Drug Levels, and Relative Biological Availability of Alternate Formulations of BMS-986460 in Healthy Adult Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA125-1018
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: BMS-986460, bioavailability, healthy adult male, crossover, SAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1: Sequence 1 (Experimental)
  Interventions: Drug: BMS-986460
- Part 1: Sequence 2 (Experimental)
  Interventions: Drug: BMS-986460
- Part 1: Sequence 3 (Experimental)
  Interventions: Drug: BMS-986460
- Part 2: Treatment A (Experimental)
  Interventions: Drug: BMS-986460
- Part 2: Treatment B (Experimental)
  Interventions: Drug: BMS-986460
- Part 2: Optional Treatment C (Experimental)
  Interventions: Drug: BMS-986460
- Part 2: Optional Treatment D (Experimental)
  Interventions: Drug: BMS-986460
- Part 2: Optional Treatment E (Experimental)
  Interventions: Drug: BMS-986460

INTERVENTIONS:
Drug: BMS-986460 — Specified dose on specified days.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, drug levels, and relative bioavailability of alternate formulations of BMS-986460 in healthy adult male participants.

ELIGIBILITY:
Inclusion Criteria

* Participants must be healthy as determined by no clinically significant deviation from normal in medical history, physical examination, vital signs, 12-lead ECGs, echocardiogram or clinical laboratory assessments, as determined by the investigator.
* Participants must have a Body mass index (BMI) between 18.0 and 35.0 kilograms/meter square (kg/m2), inclusive.
* Male participants who are sexually active with individuals of childbearing potential (IOCBP) must agree to follow instructions for methods of contraception.

Exclusion Criteria:

* Participants with prior exposure to BMS-986460 or with a prior history of heart failure, ischemic heart diseases, clinically significant cardiac arrythmias, or long QT syndrome are excluded.
* Participants with left ventricular ejection fraction (≤ 50%) at screening are excluded.
* Participants with history of anaphylactic reactions are excluded.
* Participants with current or recent (within 3 months of intervention administration) gastrointestinal disease that, in the opinion of the investigator, could affect the absorption of study intervention are excluded.
* Participants with history of Gilbert's syndrome are excluded.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AEs) | Up to approximately Day 43
Part 1: Number of Participants With Serious AEs (SAEs) | Up to approximately Day 43
Part 1: Number of Participants With Clinically Significant Physical Evaluation (PE) Findings | Up to approximately Day 21
Part 1: Number of Participants With Clinically Significant Vital Sign Abnormalities | Up to approximately Day 21
Part 1: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | Up to approximately Day 21
Part 1: Number of Participants With Clinically Significant 12-lead Electrocardiogram (ECG) Findings | Up to approximately Day 21
Part 1: Maximum Observed Plasma Concentration (Cmax) of BMS-986460 | Up to approximately Day 21
Part 1: Time of Maximum Plasma Observed Concentration (Tmax) of BMS-986460 | Up to approximately Day 21
Part 1: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC [0-T]) of BMS-986460 | Up to approximately Day 21
Part 1: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC(INF)) of BMS-986460 | Up to approximately Day 21
Part 1: Relative Bioavailability (rBA) of Alternate Formulations of BMS-986460 as Compared to Reference Formulation Based on Geometric Mean Ratio (GMR) of Cmax | Up to approximately Day 21
Part 1: rBA of Alternate Formulations of BMS-986460 as Compared to Reference Formulation Based on GMR of AUC(0-T) | Up to approximately Day 21
Part 1: rBA of Alternate Formulations of BMS-986460 as Compared to Reference Formulation Based on GMR of AUC(INF) | Up to approximately Day 21
Part 2: Number of Participants With AEs | Up to approximately Day 29
Part 2: Number of Participants With SAEs | Up to approximately Day 29
Part 2: Number of Participants With Clinically Significant PE Findings | Up to approximately Day 7
Part 2: Number of Participants With Clinically Significant Vital Sign Abnormalities | Up to approximately Day 7
Part 2: Number of Participants With Clinically Significant Laboratory Assessment Abnormalities | Up to approximately Day 7
Part 2: Number of Participants With Clinically Significant 12-lead ECG Findings | Up to approximately Day 7
Part 2: Cmax of BMS-986460 | Up to approximately Day 7
Part 2: Tmax of BMS-986460 | Up to approximately Day 7
Part 2: AUC [0-T] of BMS-986460 | Up to approximately Day 7
Part 2: AUC(INF) of BMS-986460 | Up to approximately Day 7

SECONDARY OUTCOMES:
Part 2: Pharmacokinetic (PK) Linearity of BMS-986460 Based on Cmax | Up to approximately Day 7
Part 2: PK Linearity of BMS-986460 Based on AUC(0-T) | Up to approximately Day 7
Part 2: PK Linearity of BMS-986460 Based on AUC(INF) | Up to approximately Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06877702.html